CLINICAL TRIAL: NCT01590082
Title: Phase I / II Study of the Combination of Doxycycline With Temozolomide and Ipilimumab in Patients With Metastatic Melanoma
Brief Title: Doxycycline, Temozolomide and Ipilimumab in Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Accrual slow due to alternate trials and treatment options.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-1165; NCI-2014-01836 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Results first posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Melanoma
Keywords: Melanoma; Metastatic Melanoma; Advanced melanoma; Doxycycline; Ipilimumab; Yervoy; MDX010; BMS-734016; Temozolomide; Temodar
MeSH Terms: conditions — Melanoma | interventions — Doxycycline; Ipilimumab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doxycycline, Ipilimumab, and Temozolomide (Experimental): Doxycycline to start on day -6 of Cycle 1 (1 week before Day 1 of Cycle 1 starts) twice a day until morning of Day 1 of Cycle 1. After the Day 1 of Cycle 1, participants receive first dose of Ipilimumab, and evening of same day, Temozolomide received by mouth once a day for 4 days. Doxycycline administration will continue twice daily for rest of cycle without interruption; Cycle 1 is 4 weeks of treatment. Starting Cycle 2, Doxycycline with temozolomide and ipilimumab administration start on Day 1. Each cycle is 3 weeks. 4 cycles of therapy given over a 3 month period to complete induction phase. After induction therapy, participants continue on Doxycycline.
  Interventions: Drug: Doxycycline; Drug: Ipilimumab; Drug: Temozolomide

INTERVENTIONS:
Drug: Doxycycline — Phase I Starting Dose: 200 mg by mouth twice a day on Day -6 of Cycle 1 (1 week before Day 1 of Cycle 1 starts)
  Phase II Starting Dose: Maximum Tolerated Dose (MTD) from Phase I.
Drug: Ipilimumab — Phase I and II: 3 mg by vein on Day 1 of each 21 day cycle for 4 cycles.
  Other Names: Yervoy; BMS-734016; MDX010
Drug: Temozolomide — Phase I and II: 200 mg/m2 by mouth on Days 1 - 4 of each 21 day cycle for 4 cycles.
  Other Names: Temodar

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of doxycycline that can be combined with temozolomide and ipilimumab in patients with advanced melanoma. The safety and level of effectiveness of the study drug combination will also be studied.

Doxycycline is designed to treat bacterial infection. It also blocks a protein called iNOS that is important in tumor cell growth, which may slow the growth of or kill cancer cells.

Temozolomide is designed to stop cancer cells from making new DNA (the genetic material of cells). This may stop the cancer cells from dividing into new cells.

Ipilimumab is designed to block the activity of cells that decrease the immune system's ability to fight cancer.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 5 groups of 3-6 participants will be enrolled in the Phase I portion of the study, and up to 28 participants will be enrolled in Phase II.

If you are enrolled in the Phase I portion, the dose of doxycycline you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of doxycycline. Each new group will receive a higher dose of doxycycline than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of doxycycline is found.

If you are enrolled in the Phase II portion, you will receive doxycycline at the highest or most clinically active dose that was tolerated in the Phase I portion.

All participants will receive the same dose level of temozolomide and ipilimumab.

Study Drug Administration:

You will start taking doxycycline on Day -6 of Cycle 1 (1 week before Day 1 of Cycle 1 starts) by mouth 2 times a day by itself for 1 week. You should fast (not eat or drink anything but water) for at least 2 hours before and 1 hour after you take the study drug.

After that, on Day 1 of Cycle 1, you will start taking the combination of temozolomide and ipilimumab. You will receive ipilimumab by vein over 90 minutes every 3 weeks.

On Day 1 of Cycle 1, you will start taking temozolomide by mouth with about 1 cup (8 ounces) of water on Days 1-4 of each cycle. You should fast for at least 2 hours before and 2 hours after you take the study drug.

You will continue taking doxycycline by mouth 2 times a day throughout the study.

Each study cycle is 3 weeks except the first cycle, which is 4 weeks. This is because it includes 1 week of doxycycline given by itself.

You will be given a study drug diary to record the times and doses that you take the study drugs. You should bring the diary to each study visit. You should also bring any leftover study drug with you to each study visit.

Study visits:

At every study visit, you will be asked about any drugs you may be taking, how you are feeling, and if you have had any side effects.

On Day -6 of Cycle 1:

* You will have a physical exam if not done in the past 8 days.
* Your weight and vital signs will be measured.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) will be drawn for routine tests if this was not done in the past 8 days.
* Blood (about 4 tablespoons) will be drawn for biomarker testing. Biomarkers are found in the blood and tissue and may be related to your reaction to the study drugs.

On Day 1 of Cycles 1 and 2:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 5 tablespoons) will be drawn for routine tests and biomarker testing.
* You will have an ECG.
* On Day 1 of Cycle 1, if you are in Phase II of the study, you will have a tumor biopsy performed to test if doxycycline is able to block the iNOS protein. This biopsy is optional if you are in Phase I.

On Day 8 of Cycle 1, if you are in Phase I:

* Blood (about 5 tablespoons) will be drawn for routine tests and biomarker testing.
* Your vital signs will be measured.
* Your performance status will be recorded.

On Day 15 of Cycle 1, if you are in Phase I, blood (about 5 tablespoons) will be drawn for routine tests and biomarker testing.

On Day 1 of Cycles 3 and beyond:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) will be drawn for routine tests.

Every 6 weeks (2 cycles), you will have a CT scan, an MRI scan, and/or a bone scan to check the status of the disease.

Length of Treatment:

You may continue taking doxycycline for as long as the doctor thinks it is in your best interest. You may continue receiving temozolomide and ipilimumab for up to 4 cycles.

You will no longer be able to take the study drugs if the disease gets worse, if you start having other health problems, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the end-of-treatment visit.

End-of-Treatment Visit:

Within 4 weeks after your last dose of study drugs:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 5 tablespoons) will be drawn for routine tests and biomarker testing.
* You will have an ECG.
* You will have a tumor biopsy performed to test if there is any change in the level of iNOS protein.

This is an investigational study. Temozolomide is FDA approved and commercially available to treat advanced brain tumors. It is commonly used to treat advanced melanoma but is not FDA approved for it. Ipilimumab is FDA approved and commercially available to treat advanced melanoma. Doxycycline is FDA approved and commercially available to treat various infections, but using it to treat cancer is investigational.

Up to 58 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be age >/= 18 years.
2. Patients must have histologically or cytologically confirmed diagnosis of malignant (unresectable Stage III or Stage IV) melanoma, not amenable to resection with curative intent.
3. Patients must have metastatic melanoma which has >25% of melanoma cells stained positive for iNOS expression by chemiluminescence immunoassay analyzer (CLIA)-certified immunohistochemistry assay. However, in phase I portion of the study, the requirement of >25% of melanoma cells stained positive for iNOS expression does not apply.
4. Patients must be at least 21 days since surgery, radiation therapy and 6 weeks after immunotherapy with regimens including vaccines, interferon, IL-2, etc. and fully recovered from adverse effects of these therapies.
5. Patients must have evaluable disease for response.
6. There is no limit on the number of prior therapies for Phase I portion. For Phase II portion only, patients may have received less than or equal to 1 prior chemotherapy regimen for metastatic melanoma. There is no limit on prior immunotherapies or kinase inhibitors. Patients with prior ipilimumab therapy will be excluded during the phase II portion.
7. Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or1.
8. Patient must have adequate liver and renal function as documented by the following laboratory test results within 14 days prior to starting therapy: • total bilirubin less than or equal to 1.5 x upper limit of normal (ULN); • AST (SGOT) and ALT (SGPT) less than or equal to 2.5 X ULN or less than or equal to 5 X ULN if liver metastasis is present; • serum creatinine less than or equal to 1.2 X ULN
9. Patient must have adequate bone marrow function as documented by the following laboratory test results within 14 days prior to starting therapy: • platelets greater than 100,000/mm3; • absolute neutrophil count (ANC) greater than 1500/mm3; • hemoglobin greater than 9.0 g/dL;
10. Patient must have completed any prior chemotherapy, immunotherapy, radiation therapy, biological therapy, or other investigational cancer therapy at least 4 weeks prior to starting the study drug(s) and must have recovered from all acute side effects (to Common Toxicity Criteria for Adverse Effects (CTCAE) less than Grade 1) prior to initiation of the study drug(s). Patients who were receiving mitomycin C or nitrosoureas must be 6 weeks from the last administration of chemotherapy. For a prior BRAF inhibitor, the washout period is 7 days.
11. Patient (man or woman) must agree to practice effective contraception during the entire study period, unless documentation of infertility exists, and for at least 4 weeks after the last dose of the study drug(s).
12. Patient must be willing and able to sign the informed consent form.
13. Patient must be willing and able to self-administer orally and document all doses of doxycycline ingested.
14. Patients must be willing to have iNOS expression assay test done on disease easily amenable to biopsy or suitable tissue obtained within the last 3 months.

Exclusion Criteria:

1. Patients who have received doxycycline or other tetracycline-analogs within the 4 weeks prior to the first dose of the study drug.
2. For Phase II portion only, patients with a diagnosis of ocular melanoma will be excluded.
3. Patients with an inability to swallow tablets or capsules.
4. Patients with a symptomatic malabsorptive disorder (eg, Crohn's Disease) or removal of either the terminal ileus or more than 2/3 of the small intestine.
5. Patients with active brain metastases or primary central nervous system (CNS) malignancies; patients with previously treated brain metastasis may be included, provided that no requirement for steroids and no evidence of progression for greater than or equal to 8 weeks after a local brain treatment.
6. Patients with an active second malignancy.
7. Patients who are pregnant or breastfeeding.
8. Patients with clinically significant illnesses which could compromise participation in the study, including, but not limited to:uncontrolled diabetes;active or uncontrolled infection; acute or chronic liver disease (i.e., hepatitis, cirrhosis);confirmed diagnosis of HIV infection; or, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, or uncontrolled cardiac arrhythmia.
9. Patients with history of autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sapna P. Patel, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: November 6, 2012 to March 30, 2015. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Phase I: Doxycycline + Ipilimumab + Temozolomide: Oral Doxycycline starting dose 200 mg twice a day on Day -6 of Cycle 1 (1 week before Day 1 of Cycle 1 starts), thereafter with Ipilimumab 3 mg by vein (IV) on Day 1 of each 21 day cycle for 4 cycles, oral Temozolomide 200 mg/m2 on Days 1 - 4 of each 21 day cycle for 4 cycles.
- Phase II: Oral Doxycycline 200 mg twice a day on Day -6 of Cycle 1 (1 week before Day 1 of Cycle 1 starts), thereafter with Ipilimumab 3 mg by vein (IV) on Day 1 of each 21 day cycle for 4 cycles, oral Temozolomide 200 mg/m2 on Days 1 - 4 of each 21 day cycle for 4 cycles.
Period: Overall Study
Arm/Group | Phase I: Doxycycline + Ipilimumab + Temozolomide | Phase II
Started | 11 | 1
Completed | 9 | 1
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Doxycycline + Ipilimumab + Temozolomide | Phase II | Total
Number analyzed (Participants) | 11 | 1 | 12
Age, Continuous [Median (Full Range); unit: years] | 66 [53 to 75] | 84 [84 to 84] | 67 [53 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 8 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 0 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 1 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Participant Response
Description: Number of participants with response according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria. Complete Response (CR): Disappearance all target lesions; Any pathological lymph nodes must be <10mm in short axis. Partial Response (PR): >30% decrease in sum of diameters of target lesions, reference baseline sum of diameters (e.g. percent change from baseline). Stable Disease (SD): Neither sufficient shrinkage for PR nor sufficient increase for progressive disease. Progressive Disease (PD): >20% increase in sum of diameters of target lesions, reference smallest sum of diameters recorded since treatment started (e.g. percent change from nadir, where nadir defined as smallest sum of diameters recorded since treatment start). In addition, sum must have an absolute increase from nadir of 5mm. Not Applicable (NA): No target lesions at baseline. Not Evaluable (NE): Cannot be classified by 1 of 5 preceding definitions.
Time Frame: 2 cycles, up to 7 weeks
Population: Due to early termination participants did not move to Phase 2 and no data collected.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I: Doxycycline, Ipilimumab, and Temozolomide: Oral Doxycycline starting dose 200 mg twice a day on Day -6 of Cycle 1 (1 week before Day 1 of Cycle 1 starts), thereafter with Ipilimumab 3 mg by vein (IV) on Day 1 of each 21 day cycle for 4 cycles, oral Temozolomide 200 mg/m2 on Days 1 - 4 of each 21 day cycle for 4 cycles.
Arm/Group | Phase I: Doxycycline, Ipilimumab, and Temozolomide | Phase II
Number analyzed (Participants) | 10 | 0
Participants
  Complete Response (CR) | 0 |
  Partial Response (PR) | 0 |
  Stable Disease (SD) | 3 |
  Progressive Disease (PD) | 6 |
  Not Evaluable (NE) | 1 |

ADVERSE EVENTS:
Time Frame: Adverse event evaluation Phase I: Patients will be evaluated at baseline (and/or day -6) and on days 1, 8 and 15 during cycle 1, and then on day 1 every cycle. Phase II: Patients will be evaluated ate baseline (and/or day -6) and on day 1 during cycle 1, and then on day 1 every cycle. Collection up to Cycle 5, approximately 15 weeks.
Arm/Group | Phase I: Doxycycline + Ipilimumab + Temozolomide | Phase II
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/1
Other Adverse Events (participants affected / at risk) | 9/9 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Doxycycline + Ipilimumab + Temozolomide (N=9) | Phase II (N=1)
Abdominal pain (General disorders) | 3 (4) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 5 (6) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 7 (12) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2)
Blurred vision (Eye disorders) | 3 (3) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (6) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (7) | 1 (1)
Dizziness (Nervous system disorders) | 5 (7) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Edema limbs (Musculoskeletal and connective tissue disorders) | 6 (10) | 0 (0)
Endocrine disorders - (Other (Endocrine disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 7 (13) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Infections and infestations - (Other) (Infections and infestations) | 0 (0) | 1 (2)
INR increased (Investigations) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (4) | 0 (0)
Investigations - (Other) (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (3) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (18) | 1 (1)
Pain (General disorders) | 3 (5) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 5 (7) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (7) | 0 (0)
Skin and subcutaneous tissue disorders - (Other) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (10) | 0 (0)
Weight loss (Investigations) | 5 (6) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes